CLINICAL TRIAL: NCT00329186
Title: A Randomized, Open-Label, Two-Period, Parallel Group, Crossover Study to Evaluate the Pharmacokinetics of Venlafaxine Extended-Release and DVS SR in Healthy Subjects Who Are Extensive or Poor Cytochrome P450 2D6 Substrate Metabolizers
Brief Title: Study Evaluating the Pharmacokinetics of Venlafaxine ER and Desvenlafaxine SR in Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3151A1-901
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: Healthy Subjects; Major Depressive Disorder; Depression; Cytochrome P-450 CYP2D6; Pharmacokinetics; Health
MeSH Terms: conditions — Depressive Disorder, Major; Depression

INTERVENTIONS:
Drug: desvenlafaxine SR
Drug: venlafaxine ER

SUMMARY:
The purpose of this study is to determine if the relative difference in PK between extensive metabolizers (EMs) and poor metabolizers (PMs) is the same with desvenlafaxine SR and venlafaxine ER when a single dose is administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between 18 to 55 years of age
* Healthy as determined by the investigator on the basis of medical history and physical examination, laboratory test results, vital signs, and no clinically significant abnormalities on 12-lead electrocardiogram (ECG)
* History of nonsmoker for at least 1 year

Exclusion Criteria:

* Presence or history of any disorder or significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, any severe conditions of the ears, eyes or throat (such as glaucoma or increased intraocular pressure), or psychiatric disease that may prevent the completion of the study
* Known or suspected alcohol abuse or consumption of more than 2 standard units per day within past 6 months or known or suspected abuse of prohibited drugs or other substances
* Use of any over-the-counter, prescription, hormonal therapy or investigational medications within 30 days of study day -1 until the end of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2006-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine if the relative difference in PK between EMs and PMs is the same with desvenlafaxine SR and venlafaxine ER when a single dose is administered.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Wichita, Kansas, United States

REFERENCES:
- [Derived] Preskorn S, Patroneva A, Silman H, Jiang Q, Isler JA, Burczynski ME, Ahmed S, Paul J, Nichols AI. Comparison of the pharmacokinetics of venlafaxine extended release and desvenlafaxine in extensive and poor cytochrome P450 2D6 metabolizers. J Clin Psychopharmacol. 2009 Feb;29(1):39-43. doi: 10.1097/JCP.0b013e318192e4c1. PMID 19142106